CLINICAL TRIAL: NCT04090112
Title: Comparison of Effectiveness Between the Combination of Lidocaine Sprayed at Laryngeal Inlet and on the Cuff of Endotracheal Tube Versus Intravenous Lidocaine for Reducing Cough During Extubation: A Prospective Randomized Controlled Trial
Brief Title: Comparison of Effectiveness Between the Combination of Lidocaine Sprayed at Laryngeal Inlet and on the Cuff of Endotracheal Tube Versus Intravenous Lidocaine for Reducing Cough During Extubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Pornthep Kasemsiri, Clinical Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE611394
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Reducing Cough During Extubation
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: The randomized controled trial was conducted. the investigator allocated patient into two arms. Group A received four puffs of 10% lidocaine sprayed at the cuff of ETT and four puffs at laryngeal inlet whereas Gr. B received 15 mg/kg of 2% lidocaine intravenous injection prior to extubation
Who Masked: Participant, Outcomes Assessor
Masking Description: The study based on a sequentially numbered list were prepared in the same way. Participant and outcome assessor were blined to the computer generated lists
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the study group (Group A) (Experimental): Patients received four puffs of 10% lidocaine sprayed at the cuff of ETT and four puffs at laryngeal inlet
  Interventions: Drug: 10% lidocaine sprayed
- Comparator group (Group B) (Active Comparator): Patients received 15 mg/kg of 2% lidocaine intravenous injection prior to extubation
  Interventions: Drug: 2% lidocaine intravenous

INTERVENTIONS:
Drug: 10% lidocaine sprayed — four puffs of 10% lidocaine sprayed at the cuff of ETT and four puffs at laryngeal inlet
  Other Names: 10% Xylociane
  Arms: the study group (Group A)
Drug: 2% lidocaine intravenous — 15 mg/kg of 2% lidocaine intravenous injection prior to extubation
  Other Names: 2% Xylocaine
  Arms: Comparator group (Group B)

SUMMARY:
Coughing during extubation of endotracheal tube (ETT) is a common problem that leads to poor surgical results including hemodynamic change, rebleeding at the surgical wound and wound dehiscence. Recently, lidocaine has been introduced for reducing coughing during extubation. However, data comparing routes of lidocaine application are lacking, thus, this study compared the combination of lidocaine sprayed on laryngeal inlet and cuff of ETT versus intravenous lidocaine injection for efficacy in reducing coughing

DETAILED DESCRIPTION:
A prospective randomized control trial was conduct with 164 patients. They were randomly allocated into Gr. A and B. Group A received four puffs of 10% lidocaine sprayed at the cuff of ETT and four puffs at laryngeal inlet whereas Gr. B received 15 mg/kg of 2% lidocaine intravenous injection prior to extubation. The same general anesthesia protocol was applied in all of the patients. Incidence and severity of cough during extubation was evaluated. Furthermore, incidence of 24-hour postoperative adverse events (including sore throat, dysphagia, and hoarseness) and hemodynamic response after extubation were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent elective surgery with American Society of Anesthesiologists physical status classifications of I and III

Exclusion Criteria:

* patients having body mass index more than 35 kg/m2, high risk of aspiration, chronic smokers more than ten pack-years, chronic cough or recent upper respiratory infection, suspected difficult airway, retained ETT prior surgery, surgery at oral cavity, neck and thoracic region, operative time more than 120 minutes or less than 30 minutes, and history of lidocaine allergy

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in incidence of coughing | the incidence was recorded during extubation and immediatly extubation
  Coughing event was recorded by blinded anesthesiologist

SECONDARY OUTCOMES:
Severity of coughing | the severity was recorded during extubation and immediatly extubation
  the severity of cough was recorded by blinded anesthesiologist. Coughing level severity (16) was evaluated as 0 = no cough; 1 = slight cough, cough without obvious contraction of abdomen; 2 = moderate cough, strong and sudden contraction of the abdomen lasting less than 5 seconds; 3 = severe cough, strong and sudden contraction of the abdomen sustained more than 5 seconds
Incidence of postoperative sore throat | the incidence was recorded within 24 hr after extubation
  Incidence of postoperative sore throat was recorded by two blinded anesthetist nurses . The numeric rating scale (0 = no, 10 = extreme) was used for evaluation of sore throat. If the numeric rating scale was more than 3, it was considered as a significant adverse event.
Incidence of dysphonia | the incidence was recorded within 24 hr after extubation
  Incidence of dysphonia was recorded by two blinded anesthetist nurses .
Incidence of dysphagia | the incidence was recorded within 24 hr after extubation
  Incidence of dysphagia was recorded by two blinded anesthetist nurses .

CONTACTS AND LOCATIONS:
Overall Officials: PORNTHEP KASEMSIRI, Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand

REFERENCES:
- [Result] D'Aragon F, Beaudet N, Gagnon V, Martin R, Sansoucy Y. The effects of lidocaine spray and intracuff alkalinized lidocaine on the occurrence of cough at extubation: a double-blind randomized controlled trial. Can J Anaesth. 2013 Apr;60(4):370-6. doi: 10.1007/s12630-013-9896-8. Epub 2013 Feb 1. PMID 23370978